CLINICAL TRIAL: NCT00685191
Title: HIV-1 Viral Dynamics in Subjects Initiating Raltegravir Therapy in Spain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITHACA
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: HIV Infections
Keywords: Raltegravir; HIV; dynamics; viral load; Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): HIV-1-infected subjects initiating raltegravir-including salvage therapy
  Interventions: Drug: Salvage antiretroviral therapy including raltegravir

INTERVENTIONS:
Drug: Salvage antiretroviral therapy including raltegravir — Initiation of raltegravir-including salvage antiretroviral therapy
  Other Names: RAL

SUMMARY:
The study purpose is to investigate plasma HIV-1 RNA dynamics in subjects initiating raltegravir-based salvage therapy and quantify the corresponding changes in levels of cellular HIV-1 DNA.

DETAILED DESCRIPTION:
First- and second-phase decay rates of plasma HIV-1 RNA and changes in the intracellular levels of HIV-1 proviral DNA and LTR circles will be measured in subjects starting salvage antiretroviral therapy including raltegravir in Spain.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have limited or no treatment options due to extensive antiretroviral drug resistance or drug intolerance.
* Subjects initiating raltegravir plus another fully active antiretroviral drug.

Exclusion Criteria:

* Pregnancy, or fertile women willing to be pregnant.
* Active substance abuse or major psychiatric disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-06; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Change in viral load from day 0 to 7 | 1 week

SECONDARY OUTCOMES:
Intracellular levels of HIV-1 proviral DNA and LTR circles | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet, MD,PhD, Principal Investigator — Hospital U. Germans Trias i Pujol
Locations (1):
- Hospital U. Germans Trias i Pujol, Badalona, Barcelona, Spain